CLINICAL TRIAL: NCT01263236
Title: A Phase I, Double-Blind, Placebo Controlled, Single and Multiple Oral Dose, Safety, Tolerability, and Pharmacokinetic Study of LY2940094 in Healthy Male Subjects
Brief Title: A Study of LY2940094 in Major Depressive Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BlackThorn Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 14095; I5J-MC-NOAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-12-16; First posted 2010-12-20 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Major Depressive Disorder
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — LY2940094

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY2940094 - single dose (Experimental): Single oral dose of 2-800 milligram (mg) LY2940094
  Interventions: Drug: LY2940094
- LY2940094 - multiple dose (Experimental): Daily oral dose of 2-200 mg LY2940094 for 14 days
  Interventions: Drug: LY2940094
- Placebo (Experimental): Single oral dose or daily oral dose for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2940094 — Administered orally
  Arms: LY2940094 - multiple dose; LY2940094 - single dose
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of ascending single and multiple oral doses of LY2940094 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males of any ethnic origin.
* Have a body mass index (BMI) between 19.0 and 30.0 kilogram/square meter (kg/m²), inclusive.
* Must be in good health, as determined by a medical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations.
* Have a calculated creatinine clearance of greater than 70 milliliter/minute (mL/min).
* Have venous access sufficient to allow blood sampling as per the protocol.
* Will have given their written informed consent to participate in the study and to abide by the study restrictions.

Exclusion Criteria:

* Male subjects who are not, or whose partners are not willing to use appropriate contraception from the time of the first dose until 3 months after the final dosing occasion.
* Have received any prescribed systemic or topical medication within 14 days of the first dose administration
* Have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days of the first dose administration (with the exception of vitamin/mineral supplements) unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety.
* Have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of the first dose administration
* Currently enrolled in, have completed or discontinued within the last 30 days from, a clinical trial involving an investigational product or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have donated or lost 50 to 499 milliliter (mL) of whole blood within 30 days, or more than 499 milliliter (mL) whole blood within 56 days preceding first dose administration.
* Have a significant history of drug allergy as determined by the Investigator.
* Have any clinically significant allergic disease (excluding non-active hay fever), or any known allergy to LY2940094 or excipients as determined by the Investigator.
* Have a semi-reclined blood pressure and pulse rate higher than 130/90 millimeters of mercury (mmHg) and 100 beats per minute (bpm), respectively, or lower than 90/50 millimeters of mercury (mmHg) and 40 beats per minute (bpm), respectively.
* Consume more than 28 units of alcohol per week or who have a significant history of alcoholism or drug/chemical abuse/dependence as determined by the Investigator.
* Have a positive urine drug screen or alcohol breath test result that indicates substance abuse at screening or at admission to any treatment period.
* Smoke more than 10 cigarettes or the equivalent in tobacco per day and willing to avoid smoking for durations of at least 10 hours.
* With, or with a history of, any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, hematological or other major disorders as determined by the Investigator.
* Have had a clinically significant illness within 4 weeks of the start of dose administration as determined by the Investigator.
* Have serum hepatitis, or who are carriers of the hepatitis B surface antigen (HBsAg) or hepatitis C antibody, or who have a positive result to the test for human immunodeficiency virus (HIV) antibodies.
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risk of participating in the study. In addition, subjects with the following findings will be excluded:

  * Confirmed Bazett's corrected QT (QTcB) interval greater than 450 millisecond (msec) in 2 of 3 electrocardiograms (ECGs).
  * Bundle branch blocks and other conduction abnormalities (including 2nd or 3rd degree Atrioventricular block, complete left bundle branch block, complete right bundle branch block or Wolffe-Parkinson-White Syndrome, defined as PR less than 110 milliseconds (msec),confirmed by a repeat electrocardiogram [ECG]) other than mild first-degree atrioventricular block (AV) block.
  * Irregular rhythms other than sinus arrhythmia or occasional rare supraventricular ectopic beats.
  * History of unexplained syncope.
  * Family history of unexplained syncope or sudden death due to long QT syndrome.
  * T wave configurations are not of adequate quality for assessing QTc intervals.
* Have previously completed or been withdrawn from this study.
* Taking any excluded medications that cannot be discontinued at Screening.
* Have a personal or family history of recurrent seizures or complicated febrile seizures.
* Have a history of significant brain trauma.
* Have epileptiform activity on baseline electroencephalogram (EEG).

The following exclusion criteria apply only to those subjects enrolling in the part of the study involving lumbar puncture (LP) procedures

* Have abnormalities in lumbar spine as determined by the investigator
* Have a history of clinically significant back pain and/or back injury
* Have evidence or history of significant active bleeding or coagulation disorder
* Have an allergy to lidocaine (Xylocaine®) or its derivatives
* Have medical or surgical conditions in which LP is contraindicated The following exclusion criterion applies only to those subjects enrolling in the part of the study involving alcohol interaction Have an intolerance or allergy toward alcohol (symptoms may include nausea, flushed face, vomiting, or hypotension) or who, in the opinion of the investigator, may not be able to tolerate 0.8 gram per kilogram (g/kg) alcohol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with clinically significant effects | Baseline to study completion

SECONDARY OUTCOMES:
Pharmacokinetics of LY2940094, maximal concentration (Cmax)- single dose | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 hours postdose
Pharmacokinetics of LY2940094, area under the concentration-time curve (AUC)- single dose | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 hours postdose
Pharmacokinetics of LY2940094, maximal concentration (Cmax) - multiple dose | pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12 hours postdose on day 1, predose on days 2-6, predose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 hours postdose on day 7
Pharmacokinetics of LY2940094, area under the concentration-time curve (AUC)- multiple dose | pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12 hours postdose on day 1, predose on days 2-6, predose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 hours postdose on day 7

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario, Canada